CLINICAL TRIAL: NCT05164185
Title: The Effect of Remote Ischemic Conditioning in Patients With Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017/2096-32
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Hypercholesteremia; Endothelial Dysfunction
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemia reperfusion +remote ischemic conditioning (Active Comparator): Active administration of short cykcles of ischemia.
  Interventions: Procedure: Remote ischemic conditioning
- Ischemia reperfusion +sham (Sham Comparator): Placebo experiment without remote ischemic conditioning.
  Interventions: Procedure: Remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Brief cycles of ischemia to a limb. A blood pressure cuff was placed around the right thigh and inflated to 200 mmHg for 4 cycles of 5 minutes.

SUMMARY:
There is an on-going discussion weather remote ischemic conditioning (RIC) is effective in limiting the damage of reperfusion injury in STEMI patients. The results from recent RCTs have been variable and most have not shown convincing positive results when analyzing hard endpoints. Hence, there is a great need to evaluate the impact of comorbidities on the effectiveness of RIC. Therefore, we have designed a study to evaluate the impact of hypercholesterolemia on the RIC response by evaluating ischemia-induced endothelial dysfunction.

Aim: To investigate the impact of hypercholesterolemia on the RIC response in counteracting ischemia-induced endothelial dysfunction.

DETAILED DESCRIPTION:
Study population:

We plan to include 12 poorly controlled/newly diagnosed subjects with familiar hypercholesterolemia (FH) and 12 age-matched control subjects.

Inclusion criteria (FH subjects)

* Poorly treated FH, defined as LDL-C >5.5 mmol/L.
* Age, >18 and <65 years of age.

Exclusion criteria

* Additional cardiovascular comorbidities such as diabetes mellitus, coronary artery disease, or kidney failure.
* Unwillingness to participate.
* Concurrently participating in another interventional trial.

Main exposure:

Remote ischemic conditioning, i.e. 4 cycles of 5 minutes of ischemia to the lower limb.

Comparision group:

Cross over design, patients preform the protocol twice, once with sham and once with RIC. Also a group of healthy matched controls will be recruited.

Outcome:

Change in FMD after 20 minutes of ischemia and 20 minutes of reperfusion with the exposure of either sham or RIC.

Design:

Randomized interventional cross-over.

ELIGIBILITY:
Inclusion Criteria:

* Poorly treated FH, defined as LDL-C >5.5 mmol/L.
* Age, >18 and <65 years of age.
* A age matched control-group.

Exclusion Criteria:

* Additional cardiovascular comorbidities such as diabetes mellitus, coronary artery disease, or kidney failure.
* Any condition which interfere with the outcome recording for example atrial fibrillation.
* Unwillingness to participate.
* Concurrently participating in another interventional trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Flow-mediated vasodilatation/endothelium-dependent vasodilatation | 20 min post-reperfusion
  A ultrasound based technic for evaluation of endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No